CLINICAL TRIAL: NCT05108298
Title: Improving Adolescent and Young Adult Self-Reported Data in ECOG-ACRIN Trials
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EAQ202; NCI-2021-07529 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAQ202 (Other: ECOG-ACRIN Cancer Research Group); ECOG-ACRIN-EAQ202 (Other: DCP); EAQ202 (Other: CTEP)
Record Dates: First submitted 2021-10-05; First posted 2021-11-04 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer, NOS; CNS Primary Tumor, NOS; Cervical Cancer, NOS; Colorectal Cancer, NOS; Leukemia, NOS; Lymphoma, NOS; Miscellaneous Neoplasm, NOS; Non-Rhabdomyosarcoma Soft Tissue Sarcoma, NOS; Testicular Nonseminomatous Germ Cell Tumor, NOS; Thyroid Cancer, NOS; Melanoma; Bone Cancer, NOS
MeSH Terms: conditions — Breast Neoplasms; Central Nervous System Neoplasms; Uterine Cervical Neoplasms; Colonic Neoplasms; Leukemia; Lymphoma; Pyloric Stenosis, Hypertrophic; Sarcoma; Thyroid Neoplasms; Melanoma; Bone Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Other - Patients will complete questionnaires online through EASEE-PRO. There will be a set of fixed questionnaires at each timepoint for both arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): 5 domain-specific HRQOL measures
  Interventions: Other: Questionnaires
- Control arm (Other): 5 pre-selected HRQOL measures
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Patients will complete questionnaires online through EASEE-PRO. There will be a set of fixed questionnaires at each timepoint for both arms. The patients will be asked to rank the 15 types of PROs according to their importance. The participants randomized to the choice arm will be asked to choose 5 of the 15 PROs to complete. The participants randomized to the fixed arm will be given a fixed 5 of the 15 PROs at each time point.

SUMMARY:
The purpose of this study is to evaluate feasibility and acceptability of completing PROs among AYAs randomized to Choice PRO vs Fixed PRO.

DETAILED DESCRIPTION:
Primary Aim: Conduct a pilot randomized controlled trial with AYAs to determine the feasibility and acceptability of completing PROs informed by AYAs' priorities. AYAs will be consented and randomized to select five HRQOL domains from a dashboard (Choice PRO) at each assessment period or to five standard HRQOL domains (Fixed PRO; physical function, pain, cognitive function, social support, finances) at each assessment period. AYAs will complete baseline, 1-, 3-, 6-, and 12-month assessments which will include a combination of CATs and static short forms. Feasibility will be operationalized as ≥ 75% completed PROs and ≥ 75% acceptability. Feasibility and acceptability will be compared between AYAs randomized to Choice PRO vs Fixed PRO. Adherence boosters (reminder calls, text messages) will be used to minimize missing data and evaluated as moderators.

Exploratory Aim: Solicit AYA preferences for how their PRO data should be shared with them and/or their providers. To inform future research, AYAs will be asked if and how participants want their PRO data to be used by their medical teams as well as if and how participants want their PRO data to be shared with them and their families.

The investigators anticipate PROMIS CATs will increase capacity for PRO data capture, AYAs randomized to Choice PRO, who are given the opportunity to choose which PRO domains to complete, will have less missing data. The investigators expect the majority of AYAs will want PRO feedback for themselves, their families, and their providers. Findings will promote and sustain the inclusion of PROs in clinical and supportive care trials, providing AYA's a voice and informing future patient-centered care tailored to the diverse needs of AYAs. By offering AYAs the opportunity to choose which PRO domains to complete based on relevance to their health-related quality of life, as opposed to completing domains pre-determined by the research team, the investigators raise the patient-centeredness of investigators assessment approach.

ELIGIBILITY:
Inclusion Criteria:

Patient must be ≥ 18 years and ≤ 39 years of age at registration. Patient must have a histologically confirmed diagnosis of primary cancer of any stage within 12 weeks (84 days) at registration.

Patient must have received, be currently receiving or planning to receive treatment for cancer, including surgery and/or chemotherapy and/or radiation therapy.

Patient must have an ECOG performance status 0-3. Patient must have a life expectancy >24 months. Patient must be able to complete questionnaires in English. Patient must have internet access through computer, tablet, or smartphone. Patient must have an email address. Patient must have a mobile phone able with text messaging capabilities. Patient must be able to accurately provide self-report data (e.g. per clinical judgment, cognitive function is intact).

Patient must be able to provide informed consent.

Exclusion Criteria:

Patient must not have a recurrence or second primary cancer. Patients must not have basal cell skin carcinoma.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate completion of PROs among AYAs randomized to Choice PRO vs Fixed PRO. | Feasibility at 1 month and acceptability at baseline
  Evaluate feasibility and acceptability of completing PROs among AYAs randomized to Choice PRO vs Fixed PRO.

OTHER OUTCOMES:
Evaluate AYAs' HRQOL priorities and HRQOL PRO trajectories | Through study completion, an average of 1 year
  The goal of the ranking exercise is to evaluate the importance of HRQOL domain rank choice PROs and examine their changes over time.
Access and Utilization | Assessed up to 52 months
  To evaluate access to and utilization of psychosocial and financial resources using items from the Consumer-Based Cancer Care Value Index (CCVI).
To summarize AYAs' preferences for how their PRO data should be shared with them, their families, and/or their providers. | Assessed up to 52 months
  Solicit AYAs preferences with regard to possible applications for their PRO data, including sharing PRO data with their medical teams and/or their families, and providing participants with summary feedback.

CONTACTS AND LOCATIONS:
Overall Officials: John M Salsman, PhD, Study Chair — ECOG-ACRIN Cancer Research Group
Locations (347):
- United States (347):
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Epic Care-Dublin, Dublin, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Mercy Cancer Center, Merced, California
  - Bay Area Tumor Institute, Oakland, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Beebe South Coastal Health Campus, Frankford, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Bromenn Lifecare Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Mission Cancer and Blood - Ankeny, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Mission Cancer and Blood - West Des Moines, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mission Cancer and Blood - Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Mercy Health - Paducah Medical Oncology and Hematology, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Cancer Care Specialists - Reno, Reno, Nevada
  - University of Nevada at Reno Veterans Affairs Medical Center, Reno, Nevada
  - Holy Name Hospital, Teaneck, New Jersey
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - CaroMont Health - Lincoln Cancer Center, Lincolnton, North Carolina
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Memorial Hospital, Marysville, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Mount Carmel New Albany Surgical Hospital, New Albany, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Mercy Health Sylvania Radiation Oncology Center, Toledo, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Fox Chase Cancer Center - East Norriton Hospital Outpatient Center, East Norriton, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Wellmont Medical Associates-Bristol, Bristol, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Overlake Medical Center, Bellevue, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Valley Medical Center, Renton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming

IPD SHARING:
Plan to Share IPD: No